CLINICAL TRIAL: NCT00335595
Title: Randomized, Multicenter, Phase III Study, to Evaluate the Efficacy and Safety of Bevacizumab Alone or Combined With Capecitabine and Oxaliplatin as Support Therapy After Initial Chemotherapy Treatment With Capecitabine, Oxaliplatin and Bevacizumab in Metastatic Colorectal Cancer Patients
Brief Title: Study of Bevacizumab Alone or Combined With Capecitabine and Oxaliplatin as Support Therapy in Metastatic Colorectal Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Sanofi (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-05-02; EudraCT Nº: 2005-003325-67
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; Bevacizumab; capecitabine; oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): XELOXA
  Interventions: Drug: XELOXA
- 2 (Experimental): XELOXA-A
  Interventions: Drug: XELOXA-A

INTERVENTIONS:
Drug: XELOXA — XELOXA Bevacizumab: 7,5 mg/kg, day 1 Oxaliplatino: 130 mg/m2 ; day 1 Capecitabine: 1000 mg/m2 bid, oral, day 1-14 One cycle every 3 weeks
  Arms: 1
Drug: XELOXA-A — XELOXA-A Bevacizumab: 7,5 mg/kg, day 1 Oxaliplatino: 130 mg/m2 ; day 1 Capecitabine: 1000 mg/m2 bid, oral, day 1-14 during 6 cycles followed by Bevacizumab until disease progression or premature drop out of study.
  One cycle every 3 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to compare the free time to disease progression of combination therapy with capecitabine, oxaliplatin and bevacizumab until disease progression versus capecitabine, oxaliplatin and bevacizumab for 6 cycles followed by bevacizumab until disease progression or a premature drop out of the study.

DETAILED DESCRIPTION:
The purpose of this study is to compare the free time to disease progression of combination therapy with capecitabine, oxaliplatin and bevacizumab until disease progression versus capecitabine, oxaliplatin and bevacizumab for 6 cycles followed by bevacizumab until disease progression or a premature drop out of the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent given.
* Patients who are able to understand the study request.
* Men and women > or = 18 years, not hospitalized.
* Outpatients with ECOG performance status ≤ 2.
* Histologically confirmed diagnosis of colorectal cancer (CRC) patients with metastasis.
* Presence of at least one detectable lesion in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Life expectancy of greater than 3 months.
* Men and women potentially fertile using an effective contraceptive method

Exclusion Criteria:

* Patients who have been treated with bevacizumab previously.
* Received any systemic treatment previously to treat an advanced or metastatic disease

  * Adjuvant or neoadjuvant treatment to non-metastatic disease is allowed, provided that it has been finished at least 6 months before the initial study treatment.
  * If the patient has been treated with adjuvant therapy previously, it is not allowed to be included in the study in case of disease progression during treatment or for 6 months after the end of treatment.
  * If radiotherapy has not been administered in the lesion selected for the study, previous radiotherapy is allowed, unless progression of those injuries can be documented in the radiated field, as long as the end of the treatment has been finished at least 4 weeks before study initiation.
  * Previous surgical procedure of stage IV disease is allowed.
* Previous malignancies other than adequately treated in situ carcinoma of the uterine cervix, basal or squamous cell carcinoma of the skin, or this study indication, unless there has been a disease-free interval of at least 2 years.
* History or evidence upon physical examination of central nervous system
* History of psychiatric disability judged by the investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake.
* Clinically significant cardiovascular disease (active).
* Patients who have undergone myocardial infarction or cerebrovascular accident 6 months prior to randomisation will be excluded.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome or inability to take oral medications.
* Patients subjected to allogeneic transplant and request immunotherapy.
* Bone fracture not healed, wounds or severe ulcers.
* Known hemorrhagic diathesis or coagulopathy.
* Uncontrolled and severe intercurrent infections or other severe and uncontrolled concomitant diseases.
* Moderate or severe renal impairment (creatinine clearance < 30 ml/min [calculated according to Cockroft-Gault formula] or serum creatinine ≥ 2 mg/dl or 177 μmol/l).
* Any of the following laboratory values:

  * Absolute neutrophil count (ANC) ≤ 1.5 x 10^9/l.
  * Platelet count ≤ 100 x 10^9/l.
  * Hemoglobin ≤ 9 g/dl.
  * International Normalized Ratio (INR) ≥ 1.5.
  * Total bilirubin ≥ 1.5 x upper limit of normal (ULN).
  * ALT and/or AST ≥ 2.5 x ULN or ≥ 5 x ULN (in case of hepatic metastasis).
  * Alkaline phosphatase > 2.5 x ULN or 5 x ULN (in case of hepatic metastasis), or > 10 x ULN (in case of bone metastasis).
* History of unexpected serious adverse events to fluoropyrimidine treatments or known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Patients subjected to major surgical procedure or open biopsy; or patients have had significant traumatic injuries 28 days before the initial study treatment; or patients with a major surgical procedure planned during the study period.
* Fine needle aspiration biopsy 7 days before study initiation.
* Use of full dose of oral or parenteral anticoagulants (at least 10 days before the initial study treatment) or thrombolytic agents. Low dose of warfarin is allowed, with an INR ≤ 1.5.
* Subjects requiring chronic use of high dose aspirin (> 325 mg/day) or non-steroidal anti-inflammatory treatment (those known to inhibit platelet function at doses used to treat chronic inflammatory diseases).
* Pregnant or lactating women.
* Patients with known allergy to Chinese hamster ovary cell proteins or other recombinant human or humanized antibodies; or to any excipients of bevacizumab formulation; or to any other study drugs.
* Received any investigational drug or agent/procedure, i.e. participation in another treatment trial within 30 days of randomisation.
* Evidence of another disease, metabolic malfunction, discovery in a physical examination or in a clinical laboratory test to result in reasonable suspicion of a condition or disease that contraindicates investigational medicine use or exposes the patient to high risk treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2006-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Determine the free time to disease progression | 2006-2012

SECONDARY OUTCOMES:
Overall survival | 2006-2012
Overall response rate | 2006-2012
Time to onset of response | 2006-2012
Duration of response | 2006-2012
Treatment cycles number | 2006-2012
Number of patients who need medicine dose reduction | 2006-2012
adverse events | 2006-2012
Prognostic and predictive factor of Circulating endothelial cells (CEC) and circulating tumors cells (CTC) baseline and after 3 cycle | 2006-2012
Prognostic factor of the K-Ras gene mutation | 2006-2012

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Aranda, MD; phD, Study Chair — Spanish Cooperative Group for Gastrointestinal Tumour Therapy (TTD); Eduardo Díaz-Rubio, MD; phD, Study Chair — Spanish Cooperative Group for Gastrointestinal Tumour Therapy (TTD)
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Madrid, Spain

REFERENCES:
- [Background] Sastre J, Maestro ML, Gomez-Espana A, Rivera F, Valladares M, Massuti B, Benavides M, Gallen M, Marcuello E, Abad A, Arrivi A, Fernandez-Martos C, Gonzalez E, Tabernero JM, Vidaurreta M, Aranda E, Diaz-Rubio E. Circulating tumor cell count is a prognostic factor in metastatic colorectal cancer patients receiving first-line chemotherapy plus bevacizumab: a Spanish Cooperative Group for the Treatment of Digestive Tumors study. Oncologist. 2012;17(7):947-55. doi: 10.1634/theoncologist.2012-0048. Epub 2012 May 29. PMID 22643538
- [Background] Diaz-Rubio E, Gomez-Espana A, Massuti B, Sastre J, Reboredo M, Manzano JL, Rivera F, Safont MJ, Montagut C, Gonzalez E, Benavides M, Marcuello E, Cervantes A, Martinez de Prado P, Fernandez-Martos C, Arrivi A, Bando I, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumors (TTD). Role of Kras status in patients with metastatic colorectal cancer receiving first-line chemotherapy plus bevacizumab: a TTD group cooperative study. PLoS One. 2012;7(10):e47345. doi: 10.1371/journal.pone.0047345. Epub 2012 Oct 12. PMID 23174912
- [Background] Diaz-Rubio E, Pietrantonio F, de Braud F. Continuing single-agent bevacizumab as maintenance therapy after induction XELOX (or FOLFOX) plus bevacizumab in first-line treatment of metastatic colorectal cancer. Oncologist. 2012;17(11):1426-8. doi: 10.1634/theoncologist.2012-0075. Epub 2012 Oct 16. PMID 23073991
- [Result] Diaz-Rubio E, Gomez-Espana A, Massuti B, Sastre J, Abad A, Valladares M, Rivera F, Safont MJ, Martinez de Prado P, Gallen M, Gonzalez E, Marcuello E, Benavides M, Fernandez-Martos C, Losa F, Escudero P, Arrivi A, Cervantes A, Duenas R, Lopez-Ladron A, Lacasta A, Llanos M, Tabernero JM, Anton A, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumors. First-line XELOX plus bevacizumab followed by XELOX plus bevacizumab or single-agent bevacizumab as maintenance therapy in patients with metastatic colorectal cancer: the phase III MACRO TTD study. Oncologist. 2012;17(1):15-25. doi: 10.1634/theoncologist.2011-0249. Epub 2012 Jan 10. PMID 22234633
- [Derived] Sastre J, Vidaurreta M, Gomez A, Rivera F, Massuti B, Lopez MR, Abad A, Gallen M, Benavides M, Aranda E, Rubio ED; Spanish Cooperative Group for the Treatment of Digestive Tumors. Prognostic value of the combination of circulating tumor cells plus KRAS in patients with metastatic colorectal cancer treated with chemotherapy plus bevacizumab. Clin Colorectal Cancer. 2013 Dec;12(4):280-6. doi: 10.1016/j.clcc.2013.06.001. Epub 2013 Sep 5. PMID 24012456
- See also: Related Info — http://www.ttdgroup.org